CLINICAL TRIAL: NCT02818920
Title: Pembrolizumab Prior to Surgery for Stage 1B, 2 or 3A Non-small Cell Lung Cancer (NSCLC): A Phase II Study
Brief Title: Neoadjuvant Pembrolizumab
Acronym: TOP 1501
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neal Ready MD PhD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Neal Ready MD PhD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071629
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: Pembrolizumab; Neoadjuvant; Tumor Infiltrating Lymphocytes (TILs)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab prior to and after surgery (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (prior to surgery) 200 mg IV over 30 min, days 1 & 22, two cycles; followed by surgery; followed by standard adjuvant chemotherapy (per med. oncologist) +/- radiation therapy per institutional standard of care; followed by adjuvant pembrolizumab 200 mg IV over 30 min every 21 days for 4 cycles
  -Note: Standard radiation therapy in selected patients for standard clinical indications
  Other Names: Keytruda

SUMMARY:
This multi-institutional, phase 2 clinical trial is studying two doses of pembrolizumab administered prior to surgery (neoadjuvant therapy) and 4 doses administered after surgery (adjuvant therapy) for stage IB, II or IIIA non-small cell lung cancer. Pembrolizumab is a type of immunotherapy that may enhance the ability of the immune system to fight off cancer. The study will investigate the effects of pembrolizumab on the immune system and how certain immune cells, called TILs (tumor infiltrating lymphocytes), respond to pembrolizumab. Previous studies suggest that pembrolizumab could alter the immune cells in a way that the the immune cells identify cancer cells. Pembrolizumab has been approved for the treatment of advanced lung cancer, but is investigational in this setting.

DETAILED DESCRIPTION:
The presumed mechanism of action for pembrolizumab is the removal of T lymphocyte inhibition by masking the PD-1 receptor. Our hypothesis is that the masking of the PD-1 receptor by pembrolizumab results in the activation and proliferation of T lymphocytes with specificities against tumor associated antigens (TILs). In untreated lung cancer tumors, we would expect few tumors to have TIL cells with specificities against tumor associated antigens. Based on the response rate to pembrolizumab in advanced lung cancer, we hypothesize that at least 20% of lung cancers would have TIL cells with specificities against tumor associated antigens after pembrolizumab therapy.

Studying neoadjuvant pembrolizumab therapy is an attractive strategy for studying the immunologic changes caused by PD-1 (programmed death receptor 1) checkpoint masking. Most of the immunologic activity associated with pembrolizumab occurs in the tumor and surrounding microenvironment. Evaluation of post-pembrolizumab tumor will be important to understanding factors associated with pembrolizumab activity, immune tolerance, and discovery of other targets for immune therapy. Pembrolizumab has known benefit in non-small cell lung cancer. The addition of pembrolizumab for two doses prior to surgery and four doses after surgery has the potential to confer clinical benefit. Large randomized phase 3 trials are now testing whether PD-1 checkpoint antibodies improve survival as adjuvant therapy after resection of early stage lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC.
* Clinical stage IB (>/= 3 cm per CT), Stage IIA/IIB, or Stage IIIA (N0-2) amenable to surgical resection.
* Primary tumor >/= 3 cm (for all stages entered) to make it likely that excess tumor will be available after resection.
* Patient must be deemed a surgical candidate.
* ECOG performance status of 0 or 1 (Appendix C).
* No prior chemotherapy, radiation therapy or biologic/targeted therapy for current diagnosis of lung cancer.
* Adequate Organ Function
* Age ≥18 years.
* Non-pregnant. Females of child-bearing potential (not surgically sterilized or postmenopausal [a woman who is > 45 years of age and has not had menses for greater than 1 year]) must test negative for pregnancy within 48 hours prior to any initial study procedure based on a serum pregnancy test.
* No active invasive malignancy in the past 2 years other than non-melanoma skin cancer. Cancers that are in-situ are not considered invasive.
* Signed written informed consent including HIPAA according to institutional guidelines.
* Patients must agree to research blood sampling to participate in study.
* Have measurable disease based on RECIST 1.1.
* Post-op predicted FEV1 and DLCO > 40% predicted (or per institutional standard).

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry or used an investigational device within 4 weeks of the first dose of treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Concurrent administration of any other anti-tumor therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L-1, or anti-PD-L2 agent.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Inability to comply with protocol or study procedures.
* Active infection requiring antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency etc) is not considered a form of systemic treatment. Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known additional invasive malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has had major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant disorders that in the opinion of the investigator would compromise the safety of the patient or compromise the patient's ability to complete the study.
* Has received any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 30 days before or after any dose of pembrolizumab). Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.
* Has history of myocardial infarction having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications. Patients with CAD recently treated with surgery and/or stent, if stable without symptomatic angina pectoris, active ischemia are eligible.
* Has a history of interstitial lung disease
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Prisoners or subjects who are compulsorily detained involuntarily incarcerated) for treatment of either psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Tong BC, Gu L, Wang X, Wigle DA, Phillips JD, Harpole DH Jr, Klapper JA, Sporn T, Ready NE, D'Amico TA. Perioperative outcomes of pulmonary resection after neoadjuvant pembrolizumab in patients with non-small cell lung cancer. J Thorac Cardiovasc Surg. 2022 Feb;163(2):427-436. doi: 10.1016/j.jtcvs.2021.02.099. Epub 2021 Apr 9. PMID 33985811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-five subjects consented to the study. Two subjects withdrew consent before receiving protocol treatment and three were deemed ineligible.
Period: Overall Study
Arm/Group | Pembrolizumab Prior to and After Surgery
Started | 30
Completed Surgery | 25
Received Adjuvant Therapy | 17
Completed | 12
Not Completed | 18
Not completed — Unresectable | 4
Not completed — Progressed After Neoadjuvant Therapy | 1
Not completed — Went Off Study Prior to Adjuvant Therapy | 8
Not completed — Adverse Event | 3
Not completed — Developed Other Disease | 1
Not completed — Refused Further Treatment | 1

BASELINE CHARACTERISTICS:
Population: Subjects who completed surgery.
Arm/Group | Pembrolizumab Prior to and After Surgery
Number analyzed (Participants) | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [62 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Histological Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma | 8
  Squamous cell carcinoma | 15
  Non-small cell lung cancer NOS | 2
Clinical Stage [Count of Participants; unit: Participants] — Stage IB: Tumor is 3-4 centimeters and cancer has not spread to the lymph nodes.
  Stage IIA: Tumor is 4-5 centimeters and cancer has not spread to the lymph nodes.
  Stage IIB: Tumor is < or = 5 centimeters or and cancer has spread to the lymph nodes on the same side of the chest as the primary tumor. The lymph nodes with cancer are in the lung or near the bronchus.
  Stage IIIA: Tumor is < or = 5 centimeters and cancer has spread to lymph nodes on the same side of the chest as the primary tumor. The lymph nodes with cancer are around the trachea or aorta.
  Participants
    Stage IB | 7
    Stage IIA | 6
    Stage IIB | 5
    Stage IIIA | 7
History of Smoking [Count of Participants; unit: Participants]
  Never | 3
  Current user | 4
  Quit < or = 1 month | 4
  Quit > 1 month to 1 year | 2
  Quit > 1 year | 12
ECOG (Eastern Cooperative Oncology Group) Score [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. 0 = Fully active, 1 = Restricted in physically strenuous activity but ambulatory, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities, 3 = Capable of only limited selfcare, 4 = Completely disabled, 5 = Dead.
  Participants
    0 | 14
    1 | 11
    2 | 0
    3 | 0
    4 | 0
    5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Surgical Feasibility Rate as Measured by the Number of Subjects Who Undergo Surgery Following Neoadjuvant Pembrozulimab
Description: A patient who meets the eligibility criteria, has received at least 1 dose of pembrolizumab, and undergone surgery in the window of 29-56 days after initiation of pembrolizumab is considered surgically feasible. All other situations are considered infeasible.
Time Frame: 29-56 days after initiation of pembrolizumab
Population: Subjects who completed surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Prior to and After Surgery
Number analyzed (Participants) | 25
Participants | 24

2. Other Pre Specified Outcome: Objective Response Rate
Description: The percentage of patients having a complete response or a partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Time Frame: At the end of 2 cycles of neoadjuvant pembrolizumab (29-55 days after initiation)
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Disease-free Survival (DFS)
Description: DFS is defined as the time from surgical resection to disease recurrence (first disease recurrence or death, whichever comes first) after surgery.The Kaplan-Meier estimator will be used to estimate median DFS and its confidence interval.
Time Frame: Until disease recurrence or death (up to 5 years)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Blood-based Biomarker Values
Description: Changes in levels of blood-based biomarkers before and after protocol treatment and correlated with clinical outcomes, such as objective response, overall survival, and disease-free survival.
Time Frame: Baseline (day 0), before surgery (days 29-56), 3-6 weeks after surgery, and after completion of adjuvant pembrolizumab (estimated at 10.5 months from start depending on treatment components received by patient)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Detectability of Tumor Infiltrating Lymphocytes (TILs)
Description: Percentage of patients with detectable TILs, defined as greater than or equal to 0.05% (with each value also being at least twice that of the background unstimulated control value TIL)
Time Frame: End of protocol treatment (Estimated at 10.5 months from start depending on treatment components received by patient)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Adverse Events
Description: Safety will be evaluated for all treated patients using CTCAE V 4.0.
Time Frame: End of protocol treatment (estimated at 10.5 months from start depending on treatment components received by patient)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Detectability of Circulating T Cells Specific Against TAA
Description: Proportion of patients with detectable circulating T cells specific against TAA after protocol treatment.
Time Frame: End of protocol treatment (estimated at 10.5 months from start depending on treatment components received by patient)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pathologic Response Rate
Description: Pathologic response rate for neoadjuvant pembrolizumab
Time Frame: At surgery (day 29-56)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Immunomodulatory Effects
Description: Determine if the immunomodulatory effects of neoadjuvant pembrolizumab have an impact on the suppressive mechanisms, restoring functional reactivity to important anti-tumor effects cell populations. Functional TAA-specific T cell reactivities will measured at 4 time points.
Time Frame: as for outcome 4
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Detectability of Circulating T Cells Meeting New Definition of Detectability
Description: Percentage of patients with circulating T cells meeting the new definition of detectable.
Time Frame: End of protocol treatment ((Estimated at 10.5 months from start depending on treatment components received by patient)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Gene Expression of the PD-1/PD-L1 Axis
Description: Elucidate genes associated with function and modulation of the PD-1/PD-L1 axis.
Time Frame: End of protocol treatment ((Estimated at 10.5 months from start depending on treatment components received by patient)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Correlation of Pathologic Response to the Presence of TILs
Description: A Fisher exact test will be used to evaluate the association of the presence of TILs with pathologic tumor response to neoadjuvant therapy.
Time Frame: At surgery (day 29-56)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Correlation of Pathologic Response to the Quality of TILs
Description: A Fisher exact test will be used to evaluate the association of the quality of TILs with pathologic tumor response to neoadjuvant therapy.
Time Frame: At surgery (day 29-56)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Correlation of Pathologic Response to the Quantity of TILs
Description: A Wilcoxon rank sum test will be used to test the association of the quantity of TILs and pathologic response to neoadjuvant therapy.
Time Frame: At surgery (days 29-56)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Patterns of Metastases as Measured by Frequency at Site.
Description: The Kaplan-Meier estimator will be used to estimate median DFS and its confidence interval. The frequencies of metastases by site will be tabulated
Time Frame: Until disease recurrence or death (up to 5 years)]
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 10.5 months
Description: 30 patients received neoadjuvant therapy. Among them, 25 patients underwent surgery. 17 out of those 25 patients received adjuvant therapy. Therefore, the number of patients at risk was different at different treatment phases.
Arm/Group | Pembrolizumab Prior to and After Surgery
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pembrolizumab Prior to and After Surgery (N=30)
Abdominal pain (Gastrointestinal disorders) | 1/17
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1/17
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1/17
Supraventricular tachycardia (Cardiac disorders) | 1/25
Thromboembolic event (Vascular disorders) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pembrolizumab Prior to and After Surgery (N=30)
Abdominal distension (Gastrointestinal disorders) | 1/17
Abdominal pain (Gastrointestinal disorders) | 2/17
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1/17
Anemia (Blood and lymphatic system disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 5
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Aspartate aminotransferase increased (Investigations) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3/25
Atrial fibrillation (Cardiac disorders) | 6/25
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial infection (Infections and infestations) | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/17
Chills (General disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1/17
Diarrhea (Gastrointestinal disorders) | 12
Dizziness (Nervous system disorders) | 5
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1/17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1
Edema limbs (General disorders) | 3
Endocrine disorders - Other (Endocrine disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders - Other (Eye disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 12
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 1/17
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2
General disorders and administration site conditions - Other (General disorders) | 1
Headache (Nervous system disorders) | 4
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1/17
Hemorrhoids (Gastrointestinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1/17
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 3/17
Hyperthyroidism (Endocrine disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1/17
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4/25
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Lung infection (Infections and infestations) | 2/25
Mucositis oral (Gastrointestinal disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1/17
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2/17
Nausea (Gastrointestinal disorders) | 4
Neutrophil count decreased (Investigations) | 1
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2/17
Platelet count decreased (Investigations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2/17
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 4/25
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/17
Pruritus (Skin and subcutaneous tissue disorders) | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1/17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1/17
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2/17
Scrotal infection (Infections and infestations) | 1/17
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1/17
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3
Skin induration (Skin and subcutaneous tissue disorders) | 1/17
Skin infection (Infections and infestations) | 2/25
Supraventricular tachycardia (Cardiac disorders) | 1/25
Surgical and medical procedures - Other (Surgical and medical procedures) | 1/25
Thromboembolic event (Vascular disorders) | 2/25
Tremor (Nervous system disorders) | 1/17
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2/17
Vomiting (Gastrointestinal disorders) | 1
Watering eyes (Eye disorders) | 2
Weight gain (Investigations) | 1/17
Weight loss (Investigations) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02818920/Prot_SAP_000.pdf